CLINICAL TRIAL: NCT03630146
Title: iPeer2Peer Program for Adolescents With Inflammatory Bowel Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Sara Ahola Kohut, Psychologist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1000058684
Record Dates: First submitted 2018-08-09; First posted 2018-08-14 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iPeer2Peer Mentorship (Experimental): 10 sessions of 20-30 minute Skype video calls conducted over 5-12 weeks.
  Interventions: Behavioral: iPeer2Peer program
- Waitlist Control Group (Active Comparator): The control group will receive standard care but without the iPeer2Peer program.
  Interventions: Other: Waitlist control

INTERVENTIONS:
Behavioral: iPeer2Peer program — In addition to standard care, youth in the experimental group will receive the iPeer2Peer Program. The iPeer2Peer program is a peer mentorship program that will provide modeling and reinforcement of self-management by pre-screened and trained peer mentors (young adults with IBD aged 18-25 years) who have learned to function successfully with their disease. Mentors will encourage youth to develop and engage in disease self-management skills and provide social support.
  Arms: iPeer2Peer Mentorship
Other: Waitlist control — The control group will receive standard care but without the iPeer2Peer Program.
  Arms: Waitlist Control Group

SUMMARY:
The iPeer2Peer program matches teens with Inflammatory Bowel Disease (IBD) with an older mentor who has learned to manage their IBD well and can support them emotionally and socially. This study will compare two groups of teens: those who are in the iPeer2Peer program and those in the control group (no mentor).

DETAILED DESCRIPTION:
The iPeer2Peer program matches teens with Inflammatory Bowel Disease (IBD) with an older mentor who has learned to manage their IBD well and can support them emotionally and socially. This study will compare two groups of teens: those who are in the iPeer2Peer program and those in the control group (no mentor).

The proposed trial aims to examine the impact of the iPeer2Peer program on self-management skills of youth with IBD (mentees) as well as health outcomes of peer mentors in the program. This innovative program leverages the Internet, commonly used by youth, to improve access and acceptability of self-management interventions while fostering social engagement in youth with IBD, thereby potentially improving HRQL.

ELIGIBILITY:
Inclusion Criteria:

* males and females 12-18 years old,
* gastroenterologist-diagnosed IBD,
* able to speak and read English,
* access to a computer, smartphone or tablet capable of using free Skype software (note: participants who do not have adequate Internet access will be provided with portable Internet devices),
* willing and able to complete online measures.

Exclusion Criteria:

* significant cognitive impairments or
* severe co-morbid illnesses (medical or psychiatric conditions) likely to influence HRQL assessment (e.g., psychosis, active suicidal ideation),
* participating in other peer support or self-management interventions

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-03-16 (Actual)

PRIMARY OUTCOMES:
TRANSITION-Q (measuring change) | Baseline; up to 12 weeks after baseline; 6 months post program
  14-item scale that measures self-management skills in health and healthcare in adolescents with chronic health conditions.

SECONDARY OUTCOMES:
Disease Activity Survey (measuring change) | Baseline; up to 12 weeks after baseline; 6 months post program
  21-item survey to measure disease activity and alternative resources therapies used by patients. The scale used in this study is from the Brief Pain Inventory. The scale ranges from 0 to 10 and the higher the value the worse the outcome.
IBD Self-efficacy Scale for Adolescents and Young Adults (measuring change) | Baseline; up to 12 weeks after baseline; 6 months post program
  13-item disease-specific scale to assess SE toward disease management for adolescents and young adults with IBD. Scale scores range from 1 to 5. The higher value represents a better outcome.
Brief Resiliency Scale (measuring change) | Baseline; up to 12 weeks after baseline; 6 months post program
  6-item measure that assesses an individual's ability to bounce back or recover from stress. The total range is a score from 6 to 30. A higher final score represents a better outcome.
Revised Child Anxiety and Depression Scale (measuring change) | Baseline; up to 12 weeks after baseline; 6 months post program
  25-item self-report measure of anxiety and depression characteristics. Measure includes a score for total anxiety, total depression, and total anxiety and depression. The scale ranges from a minimum score of 0 to a maximum score of 3. A higher score represents a worse outcome.
PROMIS Pediatric Item Bank v.1.0 - Peer Relationships - Short Form 8a | Baseline; up to 12 weeks after baseline; 6 months post program
  15-item measure of social health via social function and overall sociability. The scale ranges from value of 0 to 4. The higher the value the better the outcome.
IMPACT-III: A Quality of Life Questionnaire for Children with Inflammatory Bowel Disease (measuring change) | Baseline; up to 12 weeks after baseline; 6 months post program
  35-item quality of life measure specific to pediatric IBD populations. Domain scores include: bowel symptoms, systemic symptoms, emotional functioning, social functioning, body image, and treatment/interventions.
Assessment of Quality if Life (AQoL-6D) (measuring change) | Baseline; up to 12 weeks after baseline; 6 months post program
  20-item self-report measure for six separately scored dimensions and a simple global "utility" score. The scores range from 1 to 5. The higher the score the worse the outcome.
Health Services Use and Out-of-Pocket Expense Diary (measuring change) | Baseline; up to 12 weeks after baseline; 6 months post program
  53-item self-report measure to assess health service use and out of pocket expenses
Mentor Behavior Scale (measuring change) | post-intervention (approximately following 12 weeks of calls)
  15-item measure of 4 factors that affect mentor quality: structure, engagement, autonomy support, and competency support. The scale ranges in values from 1 to 5. The higher the score the higher the mentor is rated.
PROMIS Adult Profile v2.0 (measuring change) | At beginning of study and at end of study (approximately 3 years later)
  For mentors only. 29-item collection of short forms from 7 health domains: depression, anxiety, physical function, pain interference, fatigue, sleep disturbance, and ability to participate in social roles and activities. The scale is scored from 1 to 5. The higher the score the worse the outcome.
PROMIS Satisfaction with Social Roles and Activities (measuring change) | At beginning of study and at end of study (approximately 3 years later)
  For mentors only. 44-item questionnaire that measures satisfaction with one's social functioning (e.g., ability to participate in social roles and activities, and satisfaction with social roles and responsibilities) and social relationships (e.g., companionship, emotional, informational and instrumental support, and social isolation) The scale ranges from scores 1 to 5. The higher the score the better the outcome.
Chronic Disease Self-Efficacy scale (measuring change) | At beginning of study and at end of study (approximately 3 years later)
  For mentors only. 33-item measure with 10 subscales. The scale ranges from scores of 1 to 10. The higher the score the better the outcome.
  subscales are conceptually divided into 3 types of self-efficacy: 1). ability to self-management behaviors, 2) ability to manage disease in general, and 3) ability to achieve outcomes.
Mentor Interaction form | Following completion of each mentee's calls (approximately following 12 weeks of calls)
  Record of interactions with mentees

CONTACTS AND LOCATIONS:
Overall Officials: Sara Ahola Kohut, PhD, Principal Investigator — The Hospital for Sick Children
Locations (4):
- Canada (4):
  - BC Children's Hospital, Vancouver, British Columbia
  - The IWK Health Centre, Halifax, Nova Scotia
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No